CLINICAL TRIAL: NCT05906797
Title: Impact of Non-surgical Periodontal Therapy in the Improvement of Early Endothelial Dysfunction in Subjects With Periodontitis: a Randomized-controlled Clinical Trial.
Brief Title: Impact of Non-surgical Periodontal Therapy in the Improvement of Early Endothelial Dysfunction in Subjects With Periodontitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-22
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Atherosclerosis; Periodontitis
MeSH Terms: conditions — Atherosclerosis; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis (Experimental): Subjects diagnosed with periodontitis according to the most recent international guidelines and without cardiovascular diseases.
  Interventions: Procedure: Non-surgical periodontal treatment
- Healthy (No Intervention): Subjects without periodontitis and with good gingival health.

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Subgingival biofilm ultrasonic debridement
  Arms: Periodontitis

SUMMARY:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment on endothelial dysfunction parameters in subjects with periodontitis and without any cardiovascular disease.

DETAILED DESCRIPTION:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment on endothelial dysfunction parameters in subjects with periodontitis and without any cardiovascular disease.

60 patients: 30 with periodontitis and 30 with healthy controls and without periodontitis history.

All the patients are assessed for clinical, periodontal, blood and non-invasive ultrasound cardiovascular parameters. Measurements are taken before and after initial periodontal treatment in the periodontal subjects.

ELIGIBILITY:
PERIODONTITIS GROUP

Inclusion Criteria:

* Clinically diagnosed with periodontitis according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Periodontal treatment, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Cardiovascular Diseases.

HEALTHY GROUP

Inclusion Criteria:

* Clinically diagnosed with healthy periodontum withouth periodontitis history according to the EFP/AAP 2017 criteria.

Exclusion Criteria:

* Scaling, antibiotics, NSAIDs, immunosuppressants during the last 6 months.
* Pregnancy.
* Cardiovascular Diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity carotid-femoral (PWV-CF) | 8 weeks
  The speed of pulse wave propagation between carotid-femoral sites
Pulse Wave Velocity carotid-femoral (PWV-CR) | 8 weeks
  The speed of pulse wave propagation between carotid-radial sites
Carotid Intima-Media Thickness (CIMT) | 8 weeks
  The thickness of the carotid intima and media
Distensibility Coefficient (DC) | 8 weeks
  The relative change in luminal area during systole for a given pressure change (pulsed pressure), will be calculated assuming the lumen to be circular.
Advanced Glycation End products (AGEs) | 8 weeks
  A group of endogenous heterogeneous compounds that are constantly formed under physiological conditions with prooxidant and cytotoxic properties. Measurements are performed by fluorescence spectroscopy technique.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: No